CLINICAL TRIAL: NCT00629850
Title: Concurrent Respiratory Resistance Training and Changes in Respiratory Muscle Strength and Sleep Quality in Persons With Spinal Cord Injury
Brief Title: Respiratory Resistance Training on Sleep Quality in Persons With Spinal Cord Injury
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: unable to recruit participants.
Sponsor: Texas State University, San Marcos (Other)
Responsible Party: Principal Investigator, Chris Russian, Principal Investigator, Texas State University, San Marcos
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TexasState 2008-29541; IRB# 2008-29541 (Other: Texas State University IRB)
Record Dates: First submitted 2008-02-25; First posted 2008-03-06 (Estimated); Results first posted 2011-08-18 (Estimated); Last update posted 2019-05-08 (Actual); Status verified 2019-04

CONDITIONS: Spinal Cord Injury
Keywords: spinal cord injury; respiratory muscle training; sleep quality
MeSH Terms: conditions — Spinal Cord Injuries; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Powerlung Performer (Experimental): The arm will receive the lung trainer device to use for 10 weeks
  Interventions: Device: Powerlung Performer
- Control (No Intervention): Control. This arm will not receive any device

INTERVENTIONS:
Device: Powerlung Performer — Inspiratory/Expiratory muscle trainer
  Other Names: Respiratory resistance trainer
  Arms: Powerlung Performer

SUMMARY:
The purpose of this study is to determine if the use of a respiratory resistance trainer will increase respiratory muscle strength, improve sleep quality and improve quality of life in individuals with spinal cord injury.

Hypothesis: Use of the respiratory resistance trainer will improve respiratory muscle strength, improve sleep quality, and improve quality of life among individuals with spinal cord injury.

DETAILED DESCRIPTION:
Individuals with spinal cord injury experience varying degrees of reduced muscle function. Those individuals with high level spinal cord injury, cervical region, may experience reduced diaphragm function. This reduction in function may affect daytime activities as well as sleep quality. Sleep quality in people with spinal cord injury is considered to be worse than sleep quality in the general population. The use of respiratory resistance training devices has been shown to increase muscle strength in people with spinal cord injury. There have been not studies to document potential improvements in sleep quality among individuals with spinal cord injury following respiratory resistance training.

ELIGIBILITY:
Inclusion Criteria:

* tetraplegia
* quadriplegia

Exclusion Criteria:

* NA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2008-02; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Lloyd, Ph.D., Study Chair — Texas State University, San Marcos
Locations (1):
- Texas State University-San Marcos, San Marcos, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Powerlung Trainer Device: The device was used twice a day. Each use consisted of two sets of 10 breaths for each set.
- Control: This arm of the study will not receive the device.
Period: Overall Study
Arm/Group | Powerlung Trainer Device | Control
Started | 1 | 0
Completed | 1 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: This was a single subject case study. No control subjects.
Groups:
- Total: Total of all reporting groups
Arm/Group | Powerlung Trainer Device | Control | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 1
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Improvement in Sleep Quality.
Description: Improvement in sleep quality as defined by: less fragmented sleep, lower apnea hypopnea index (AHI), respiratory disturbance index (RDI) after device use.
Time Frame: 10 weeks
Population: There was only one participant completing the study. No analyses performed.
Arm/Group | Powerlung Trainer Device | Control
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Change in Maximum Voluntary Ventilation Using Pulmonary Function Device
Description: Pulmonary function device measures flow rate in liters per minute over a period of at least 12 seconds.
Time Frame: 10 weeks
Population: there was only one participant completing this study. No analyses performed.
Arm/Group | Powerlung Trainer Device | Control
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Change in Negative Inspiratory Force Using a Pressure Manometer
Time Frame: 10 weeks
Population: there was only one participant completing this study. No analyses performed.
Arm/Group | Powerlung Trainer Device | Control
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 8 weeks of data collection
Description: Other adverse events.
Arm/Group | Powerlung Trainer Device | Control
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 0/1 | 0/0

LIMITATIONS AND CAVEATS:
Unable to recruit subjects for the study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes